CLINICAL TRIAL: NCT04545723
Title: The Effect of a Case-finding App on the Detection Rate of Atrial Fibrillation Compared with Opportunistic Screening in Primary Care Patients: Protocol for a Cluster Randomized Trial
Brief Title: The Effect of a Case-finding App on the Detection Rate of Atrial Fibrillation in Primary Care Patients
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Insufficient amount of recruited practices due to workload and COVID19.
Sponsor: KU Leuven (Other)
Collaborators: Qompium NV (Industry)
Responsible Party: Principal Investigator, Bert Vaes, Professor, KU Leuven
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: B3222020000036
Record Dates: First submitted 2020-09-04; First posted 2020-09-11 (Actual); Last update posted 2024-09-20 (Actual); Status verified 2024-09

CONDITIONS: Atrial Fibrillation Paroxysmal
Keywords: atrial fibrillation; screening; FibriCheck; case finding
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control group (No Intervention): In every cluster designated as a control group, patients aged 65 or older will be selected according to the inclusion criteria. The difference here is that patients will be given the standard opportunistic screening instead: pulse palpation and a 12-lead ECG when an irregular rhythm is found. This is current best practice.
- Intervention group (Active Comparator): In every cluster designated as an intervention group, patients aged 65 or older will be selected according to the inclusion criteria. Within this group, high-risk patients will be identified using the CHARGE-AF score, and will be prescribed the FibriCheck® app.
  Interventions: Device: FibriCheck

INTERVENTIONS:
Device: FibriCheck — FibriCheck is a smartphone application that measures hearth rhythm using the phone's built-in camera. It is able to detect aberrant rhythms, such as atrial fibrillation.
  Arms: Intervention group

SUMMARY:
Atrial fibrillation is a cardiac arrhythmia commonly encountered in a primary care setting. Current screening is limited to pulse palpation and ECG confirmation when an irregular pulse is found. Paroxysmal atrial fibrillation will, however, still be difficult to pick up. With the advent of smartphones, screening could be more cost-efficient by making use of simple applications, lowering the need for intensive screening to discover (paroxysmal) atrial fibrillation.

This cluster randomized trial will examine the effect of using a smartphone-based application such as FibriCheck® on the detection rate of atrial fibrillation in a Flemish general practice population. This study will be conducted in 22 primary care practices across the Flanders region of Belgium and will last 12 months. Patients above 65 years of age will be divided in control and intervention groups on the practice level. The control group will be subjected to standard opportunistic screening only, while the intervention group will be prescribed the FibriCheck® app on top of this opportunistic screening. The difference in detection rate between control and intervention groups will be calculated at the end of the study.

The investigators will use the online platform INTEGO for pseudonymized data collection and analysis, and risk calculation.

Smartphone applications might offer a way to cost-effectively screen for (paroxysmal) atrial fibrillation in a primary care setting. This could open the door for the update of future screening guidelines.

ELIGIBILITY:
Inclusion Criteria:

1. The patient is 65 years or older.
2. The patient has an electronic medical record (EMR) in the practice. This EMR contains all the patient information, for instance regarding medical history and medication and is managed by the general practitioner.
3. If the patient will be prescribed the FibriCheck® app, he/she signs the relevant patient consent form

Exclusion Criteria:

1. The patient has already been diagnosed with AF.
2. The patient is already under anticoagulant therapy.
3. The patient has a pacemaker. Active pacing during measurements influences the results obtained with the FibriCheck® app (26).
4. The patient is unable to use the FibriCheck® application independently due to cognitive disorders, functional limitations, visual impairments…

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-10 (Estimated); Primary Completion 2024-11 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Detection rate of AF in patients 65 years and older | 4 weeks for each participant
  The detection rate of AF in both the control and intervention group will be calculated after 4 weeks. A significant difference in both groups will be noted. Compared with previous studies of similar design (32-34), we will realistically assume a 2-fold increase in the detection rate of AF in the intervention group to be significant.

SECONDARY OUTCOMES:
Thromboembolic complications | 12 months
  We will track incidence of transient ischemic attack or ischemic stroke during the study period, in addition to the eventual difference between both study populations.
Death | 12 months
  We will keep track of all-cause mortality during the study period, as well as difference in mortality between control and intervention populations.
Compliance | 12 months
  We will keep track of patient compliance during the study period (e.g. minimum number of measurements with FibriCheck®).

CONTACTS AND LOCATIONS:
Overall Officials: Simon G Beerten, MD, MSc, Principal Investigator — KU Leuven; Tine Proesmans, MSc, Principal Investigator — Qompium NV; Bert Vaes, MD, PhD, Principal Investigator — KU Leuven

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data will be available upon reasonable request. The trial's dataset will be held at the University of Leuven, Belgium, and can be shared upon contacting the principal investigator.

REFERENCES:
- [Derived] Beerten SG, Proesmans T, Vaes B. The effect of a case-finding app on the detection rate of atrial fibrillation compared with opportunistic screening in primary care patients: protocol for a cluster randomized trial. Trials. 2021 Aug 9;22(1):525. doi: 10.1186/s13063-021-05497-x. PMID 34372905